CLINICAL TRIAL: NCT03947853
Title: THETIS: Non-interventional, Multicenter Clinical Study to Evaluate the Predictive Value of the Heart Failure Questionnaire (HF-Q) for the Occurrence of Μajor Αdverse Cardiovascular Events (MACE) According to New York Heart Association Functional Classification (NYHA) in Patients With Symptomatic Heart Failure
Brief Title: Clinical Study to Evaluate the Predictive Value of the Heart Failure Questionnaire (HF-Q) for the Occurrence of Μajor Αdverse Cardiovascular Events (MACE) in Patients With Symptomatic Heart Failure
Acronym: THETIS
Status: Withdrawn | Type: Observational
Why Stopped: No active recruitment
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-IVBR-EL-95
Record Dates: First submitted 2019-05-10; First posted 2019-05-13 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2019-05

CONDITIONS: Heart Failure; Heart Failure NYHA Class III; Heart Failure NYHA Class II; Heart Failure NYHA Class IV
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiac Heart Failure Questionnaire HF-Q) to assess the severity of the symptoms of Heart Failure. In this study, modified and translated, the "four-point" questionnaire by Severo and his associates - Heart Failure Questionnaire HF-Q, is used. The HF-Q Heart Failure Questionnaire consists of four closed questions: the first with four possible answers and the other three questions with the possibility of three simple-choice answers.

DETAILED DESCRIPTION:
An important new element in recent guidelines is the recommendation to prevent the onset of heart failure syndrome and / or delay its progression. The degree of patient functional limitation is determined using the New York Heart Association (NYHA) classification, which in combination with the left ventricular ejection fraction is the main criterion for all clinical studies in HF.

Specifically, NYHA's functional classification is used to describe the severity of symptoms and exercise tolerance and includes 4 classes (I-IV) :

Class I: Unbound in physical activity. Conventional physical activity does not cause fatigue, palpitations or shortness of breath.

Class II: Mild limitation to physical activity. No symptoms in the calm, but ordinary physical activity causes fatigue, palpitations or shortness of breath.

Class III: Serious restriction to physical activity. No symptoms in the calm, but even mild physical activity causes fatigue, palpitations or shortness of breath.

Class IV: Inability to perform any physical activity without discomfort. Symptoms and seclusion. Strengthening the discomfort in any physical activity.

The study evaluates the predictive capacity of the Cardiac Deficiency Questionnaire (HF-Q) for the occurrence of Adverse Cardiovascular Stroke (MACE) according to the New York Heart Association (NYHA) Functional Classification of Heart Failure in patients with symptomatic Heart Failure .

This type of approach may be useful in the reproducibility of the results and the validity of the NYHA classification system, since the severity of the heart failure symptoms is recorded on the basis of the patient's own perception.

The term MACE or "Major Unwanted Cardiovascular Syndromes" is undoubtedly the most common and complex endpoint in cardiology research. Historically, the term MACE appears to be used in the mid-1990s with its use being mainly limited to the intra-muscular complications associated with transcutaneous coronary interventions (PCIs). Despite the widespread use of the term in clinical trials, the definitions of MACE may differ, which makes it difficult to compare similar studies.

The so-called "classic 3-point MACE" is defined based on the following17:

* Cardiovascular Death
* Myocardial infarction
* Cerebral Episode (Ischemic or Haemorrhagic) In general, MACE terminology is a complex clinical event and includes endpoints that reflect both safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with symptomatic Heart Failure NYHA≥2
* Patients who have fully understood the procedures of the study and have signed an informed consent form.

Exclusion Criteria:

* Patients with asymptomatic heart failure (NYHA = 1)
* Patients with severe motor impairment / mobility impairment (neurological diseases, muscular diseases, severe anemia, previous mobility stroke, severe malignancy, end-stage COPD)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with symptomatic Heart Failure NYHA≥2
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Heart Failure Questionnaire (HF-Q) | 6 months
  HF-Q rating vs NYHA classification
Major Adverse Cardiovascular Events (MACEs) | 6 months
  Number of MACEs occured during the study

REFERENCES:
- [Background] Mosterd A, Hoes AW. Clinical epidemiology of heart failure. Heart. 2007 Sep;93(9):1137-46. doi: 10.1136/hrt.2003.025270. PMID 17699180
- [Background] Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Judd SE, Kissela BM, Lackland DT, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Willey JZ, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2015 update: a report from the American Heart Association. Circulation. 2015 Jan 27;131(4):e29-322. doi: 10.1161/CIR.0000000000000152. Epub 2014 Dec 17. No abstract available. PMID 25520374
- [Background] Mant J, Doust J, Roalfe A, Barton P, Cowie MR, Glasziou P, Mant D, McManus RJ, Holder R, Deeks J, Fletcher K, Qume M, Sohanpal S, Sanders S, Hobbs FD. Systematic review and individual patient data meta-analysis of diagnosis of heart failure, with modelling of implications of different diagnostic strategies in primary care. Health Technol Assess. 2009 Jul;13(32):1-207, iii. doi: 10.3310/hta13320. PMID 19586584
- [Background] Mentz RJ, Cotter G, Cleland JG, Stevens SR, Chiswell K, Davison BA, Teerlink JR, Metra M, Voors AA, Grinfeld L, Ruda M, Mareev V, Lotan C, Bloomfield DM, Fiuzat M, Givertz MM, Ponikowski P, Massie BM, O'Connor CM. International differences in clinical characteristics, management, and outcomes in acute heart failure patients: better short-term outcomes in patients enrolled in Eastern Europe and Russia in the PROTECT trial. Eur J Heart Fail. 2014 Jun;16(6):614-24. doi: 10.1002/ejhf.92. Epub 2014 Apr 25. PMID 24771609
- [Background] Follath F, Yilmaz MB, Delgado JF, Parissis JT, Porcher R, Gayat E, Burrows N, McLean A, Vilas-Boas F, Mebazaa A. Clinical presentation, management and outcomes in the Acute Heart Failure Global Survey of Standard Treatment (ALARM-HF). Intensive Care Med. 2011 Apr;37(4):619-26. doi: 10.1007/s00134-010-2113-0. Epub 2011 Jan 6. PMID 21210078
- [Background] Clinical guideline Published: 8 October 2014 , nice.org.uk/guidance/cg187, Acute heart failure: diagnosis and management.
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Tsioufis C, Iliakis P, Kasiakogias A, Konstantinidis D, Lovic D, Petras D, Doumas M, Tsiamis E, Papademetriou V, Tousoulis D. Non-pharmacological Modulation of the Autonomic Nervous System for Heart Failure Treatment: Where do We Stand? Curr Vasc Pharmacol. 2017;16(1):30-43. doi: 10.2174/1570161115666170428124756. PMID 28462724
- [Background] NHFA CSANZ Heart Failure Guidelines Working Group; Atherton JJ, Sindone A, De Pasquale CG, Driscoll A, MacDonald PS, Hopper I, Kistler PM, Briffa T, Wong J, Abhayaratna W, Thomas L, Audehm R, Newton P, O'Loughlin J, Branagan M, Connell C. National Heart Foundation of Australia and Cardiac Society of Australia and New Zealand: Guidelines for the Prevention, Detection, and Management of Heart Failure in Australia 2018. Heart Lung Circ. 2018 Oct;27(10):1123-1208. doi: 10.1016/j.hlc.2018.06.1042. No abstract available. PMID 30077227
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Colvin MM, Drazner MH, Filippatos GS, Fonarow GC, Givertz MM, Hollenberg SM, Lindenfeld J, Masoudi FA, McBride PE, Peterson PN, Stevenson LW, Westlake C. 2017 ACC/AHA/HFSA Focused Update of the 2013 ACCF/AHA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Failure Society of America. J Am Coll Cardiol. 2017 Aug 8;70(6):776-803. doi: 10.1016/j.jacc.2017.04.025. Epub 2017 Apr 28. No abstract available. PMID 28461007
- [Background] Raphael C, Briscoe C, Davies J, Ian Whinnett Z, Manisty C, Sutton R, Mayet J, Francis DP. Limitations of the New York Heart Association functional classification system and self-reported walking distances in chronic heart failure. Heart. 2007 Apr;93(4):476-82. doi: 10.1136/hrt.2006.089656. Epub 2006 Sep 27. PMID 17005715
- [Background] Sandra L. Carroll et al., A Comparison of the NYHA Classification and the Duke Treadmill Score in Patients with Cardiovascular Disease, Open Journal of Nursing, 2014, 4, 774-783, SciRes. http://www.scirp.org/journal/ojn, http://dx.doi.org/10.4236/ojn.2014.411083.
- [Background] Severo M, Gaio R, Lourenco P, Alvelos M, Bettencourt P, Azevedo A. Indirect calibration between clinical observers - application to the New York Heart Association functional classification system. BMC Res Notes. 2011 Aug 3;4:276. doi: 10.1186/1756-0500-4-276. PMID 21813014
- [Background] Kip KE, Hollabaugh K, Marroquin OC, Williams DO. The problem with composite end points in cardiovascular studies: the story of major adverse cardiac events and percutaneous coronary intervention. J Am Coll Cardiol. 2008 Feb 19;51(7):701-7. doi: 10.1016/j.jacc.2007.10.034. PMID 18279733
- [Background] World Medical Association.. World Medical Association Declaration of Helsinki. Ethical principles for medical research involving human subjects. Bull World Health Organ. 2001;79(4):373-4. Epub 2003 Jul 2. No abstract available. PMID 11357217